CLINICAL TRIAL: NCT04706429
Title: A Randomised, Double-blind, Placebo-controlled, Phase 2 Evaluation of the Efficacy and Mechanism of Trientine in Patients With Hypertrophic Cardiomyopathy
Brief Title: The Efficacy and Mechanism of Trientine in Patients With Hypertrophic Cardiomyopathy
Acronym: TEMPEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Manchester (Other); University of Liverpool (Other); Univar BV (Industry); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B00844; 2020-002242-17 (EudraCT Number); ISRCTN57145331 (Registry Identifier: ISRCTN); NIHR127575 (Other Grant/Funding Number: NIHR EME Programme)
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Trientine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trientine (Active Comparator): Trientine dihydrochloride 1200 mg per day. This shall be taken orally as two Cufence 200mg hard capsules two times per day. The IMP will be dispensed to participants every 13 weeks for the duration of the study period (52 weeks).
  Interventions: Drug: Trientine
- Placebo (Placebo Comparator): The placebo shall be taken orally as two capsules two times per day. This will be dispensed to participants every 13 weeks for the duration of the study period (52 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trientine — Trientine dihydrochloride is a white to pale yellow crystalline hygroscopic powder.
  Other Names: Cufence
  Arms: Trientine
Drug: Placebo — Placebo capsule, manufactured with the exact components of the trientine capsules, without the active ingredient / investigational medicinal product.
  Arms: Placebo

SUMMARY:
This research study has been designed to test whether a drug called trientine dihydrochloride (also called Cufence) reduces heart muscle thickening, improves exercise capacity, improves heart function and reduces abnormal heart rhythms in patients with hypertrophic cardiomyopathy (HCM). The study is also assessing how trientine works in HCM. Participants will be prescribed either trientine or placebo, for a period of 12 months.

DETAILED DESCRIPTION:
HCM is the most common inherited cardiovascular disorder. It is characterised by left ventricular (LV) myocardial hypertrophy and fibrosis. Patients can experience symptoms of effort intolerance, progressive heart failure and abnormal heart rhythms. There are currently no treatments that alter the natural history of HCM. Patients and the cardiovascular field have identified a "critical need" for clinical studies of drug therapies that target HCM pathophysiological mechanisms.

Trientine dihydrochloride is a copper-chelating agent licensed for Wilson disease, a genetic disorder of copper excretion, in which patients exhibit a cardiac phenotype that mimics HCM. Proof of concept has been established through an MRC-funded study to suggest that use of trientine may also be beneficial in HCM.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age 18-75 inclusive.
3. Hypertrophic cardiomyopathy (HCM), as defined by the European Society of Cardiology HCM guidelines as: "a wall thickness ≥15 mm in one or more LV myocardial segments that is not explained solely by loading conditions". The same definition is applied to first-degree relatives of patients with HCM i.e. all participants are required to have a LV wall thickness ≥15 mm. Wall thickness is as measured on the most recent cardiovascular magnetic resonance (CMR) scan performed prior to the baseline visit. If CMR has not been performed previously, wall thickness measurement should be taken from the most recent echocardiogram performed prior to the baseline visit. (It is recognised that in the European Society of Cardiology guidelines a clinical diagnosis of HCM in first-degree relatives requires a wall thickness that is less than this value, however ≥15 mm is applied here in order to ensure that all participants have an unequivocal phenotype).
4. New York Heart Association class I, II or III at the most recent clinical assessment performed prior to the baseline visit.

Exclusion Criteria:

1. Previous or planned septal reduction therapy.
2. Previously documented myocardial infarction or severe coronary artery disease.
3. Uncontrolled hypertension, defined as a systolic blood pressure of >180mmHg or a diastolic blood pressure of > 100mmHg at Visit 1.
4. Known LV EF < 50%, as measured on the most recent CMR scan performed prior to the baseline visit. If CMR has not been performed previously, the most recent echocardiogram performed prior to the baseline visit should be used.
5. Previously documented persistent atrial fibrillation.
6. Anaemia, defined as haemoglobin being below the local site normal reference range, at Visit 1.
7. Iron deficiency, defined as serum iron being below the local site normal reference range, at Visit 1.
8. Copper deficiency, defined as serum copper being below the normal reference range, at Visit 1.
9. Pacemaker or implantable cardioverter defibrillator.
10. Known severe valvular heart disease, as demonstrated on the most recent heart imaging performed prior to the baseline visit.
11. Previously documented other cardiomyopathic cause of myocardial hypertrophy (e.g. amyloidosis, Fabry disease, mitochondrial disease).
12. History of hypersensitivity to any of the components of the investigational medicinal product (IMP).
13. Known contraindication to MRI scanning.
14. Pregnancy, lactation or planning pregnancy. Women of childbearing capacity are required to have a negative serum pregnancy test before treatment, must agree to pregnancy tests at study visits as defined in the Section 8 and must agree to maintain highly effective contraception as defined in Section 8 during the study.
15. Any medical condition, which in the opinion of the Investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass indexed to body surface area (LVMi) | 12 months
  Change in LVMi (g/m2), measured using CMR, from baseline to week 52.

SECONDARY OUTCOMES:
Urine copper excretion | 12 months
  Cumulative urine copper excretion, measured using urinary copper, assessed from baseline to weeks 13, 26, 39 and 52.
Exercise capacity | 12 months
  Change in exercise capacity, measured using cardiopulmonary exercise testing (CPET), assessed from baseline to week 52.
Number of non-sinus supraventricular heart beats, presence and amount of atrial fibrillation, number of ventricular-origin beats and presence and amount of non-sustained ventricular tachycardia | 12 months
  Change in number of non-sinus supraventricular heart beats, presence and amount of atrial fibrillation, number of ventricular-origin beats and presence and amount of non-sustained ventricular tachycardia, in 24 hours, measured using ambulatory heart monitoring, assessed from baseline to week 52.
Circulating high sensitivity troponin | 12 months
  Change in circulating high sensitivity troponin, assessed from baseline to week 52.
LV global longitudinal strain, wall thickness, mass, volumes and ejection fraction (EF) | 12 months
  Change in LV global longitudinal strain, wall thickness, mass, volumes and ejection fraction (EF) measured using CMR, assessed from baseline to week 52.
Peak left ventricular outflow | 12 months
  Change in peak left ventricular outflow tract gradient, measured using CMR, assessed from baseline to week 52.
Atrial volume and function | 12 months
  Change in atrial volume and function, measured using CMR, assessed from baseline to week 52.

OTHER OUTCOMES:
LV myocardial cellular mass | 12 months
  Change in LV myocardial cellular mass, measured using CMR, from baseline to week 52.
LV myocardial extracellular mass | 12 months
  Change in LV myocardial extracellular mass, measured using CMR, from baseline to week 52.
LV myocardial extracellular volume | 12 months
  Change in LV myocardial extracellular volume, measured using CMR, from baseline to week 52.
LV late gadolinium enhancement | 12 months
  Change in LV late gadolinium enhancement, measured using CMR, from baseline to week 52.
PCr/ATP ratio | 12 months
  Change in PCr/ATP ratio, measured using 31P MRS (sub-group), from baseline to week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Miller, Principal Investigator — Manchester University NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - NHS Grampian, Aberdeen
  - University Hospitals of Leicester NHS Foundation Trust, Leicester
  - Liverpool Heart and Chester Hospital NHS Foundation Trust, Liverpool
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farrant J, Dodd S, Vaughan C, Reid A, Schmitt M, Garratt C, Akhtar M, Mahmod M, Neubauer S, Cooper RM, Prasad SK, Singh A, Valkovic L, Raman B, Ashkir Z, Clayton D, Baroja O, Duran B, Spowart C, Bedson E, Naish JH, Harrington C, Miller CA; TEMPEST investigators. Rationale and design of a randomised trial of trientine in patients with hypertrophic cardiomyopathy. Heart. 2023 Jul 12;109(15):1175-1182. doi: 10.1136/heartjnl-2022-322271. PMID 37137675